CLINICAL TRIAL: NCT01598220
Title: Efficacy Study of a Computer Cognitive Remediation Program in Patients With Schizophrenia
Brief Title: Computer Assisted Cognitive Remediation Program in Schizophrenia
Acronym: CACREPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gemma Garrido García (Other)
Responsible Party: Sponsor-Investigator, Gemma Garrido García, Efficacy study of a computer cognitive remediation program in patients with schizophrenia, Consorci Sanitari de Terrassa
Organization: Consorci Sanitari de Terrassa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CACR-2012-MT
Record Dates: First submitted 2012-04-03; First posted 2012-05-15 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Schizophrenia
Keywords: schizophrenia; cognitive remediation therapy; cognition; quality of life
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computer-assisted cognitive remediation therapy (Experimental)
  Interventions: Behavioral: Computer-assisted cognitive remediation therapy
- attentional task (Placebo Comparator)
  Interventions: Other: attentional task

INTERVENTIONS:
Behavioral: Computer-assisted cognitive remediation therapy — Comparison of two groups:
  The experimental group performs 48 sessions of computer exercices designed to remedy cognitive domains(attention, speed of processing, working memory,reasoning and problem solving) frequently affected in schizophrenia.
  The intervention has a period 6 months , two sessions a week. All exercises provided a visual or verbal feedback to immediately terminate the execution.In addition to, the therapist after the sessions interactively explain the results and the strategies employed by the patient.
  Other Names: cognitive remediation therapy
  Arms: Computer-assisted cognitive remediation therapy
Other: attentional task — The Control group performs 48 sessions of watching videos and answer questions about these videos, in a period of 6 months , two sessions a week.
  Arms: attentional task

SUMMARY:
The purpose of this study is to determine whether computer-assisted cognitive remediation therapy is effective in the treatment of cognitive deficits in schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia can be considered a chronic illness that affects all aspects of daily life. Cognitive deficits seems to play a key role that interferes directly in the functional adaptation.

Cognitive remediation therapy (CRT) emerges as a psychological intervention that target cognitive impairment. But, the use of computerized or papel an pencil procedures for remediation cognitive deficits remains controversial. Nonetheless, computer tasks offer a number of advantages compared to those of paper and pencil. The most noteworthy advantages are to enhance patient's motivation just because the sensory variety that the exercises presented or the possibility to provide immediate feedback. Furthermore, the possibility to present custom-tailored and adapted tasks taking into accounts the patients deficits and their evolution in the process of the psychological therapy is another important feature of computer-assisted cognitive remediation therapy.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV (APA, 1994)criteria for schizophrenia disorder
* Estimated IQ of 85 or superior by Vocabulary subtest, Wechsler Adult Intelligence Scale-III (WAIS-III)
* Patients were considered sufficiently stable if they had a Global Assessment of Functioning Scale (GAF)score of 40 or superior and they maintained a stable dose and type of psychiatric medication for at least 1 moth prior to inclusion.

Exclusion Criteria:

* Non presence of cognitive impairment confirmed by neurocognitive assessment
* Traumatic brain injury or history of neurologic illness.
* Electroconvulsive therapy in the last year.
* Psychiatric comorbidity.
* Plan to change medication during the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2002-09; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Change in neurocognitive outcomes | Change from Baseline in neurocognitive measures up to the end of intervention at 6 months
  Attention:Continuous Performance TestII(CPT II)d'índex, Psychomotor Speed:Symbol Digit Modalities Test (SDMT; Smith, 1973,2002). Phonemic fluency FAS test (Benton & Hamsher 1976, 1989).Working Memory: Subtest Letter-Number Sequencing (WAIS-III):Verbal Learning:California Verbal Learning Test (CVLT, Delis et al 2000)short- term and long-term free recall.Executive function: Wisconsing Card Sorting Test(WCST; R.Heaton computer version CV3) categories and perseverations, Stroop test ( Stroop Color and Word Test; Stroop,1935; Golden,1994) , Matrix Reasoning (Adult Intelligence Scale-III ;WAIS-III).

SECONDARY OUTCOMES:
Change in functional outcomes | Change from Baseline in functional measures up to the end of intervention at 6 months
  The Heinrichs -Carpenter Quality of life Scale.(QLS, Heinrichs,1982; Spanish version Rodríguez et al.1995).QLS are divided in four subscales socialactivity, interpersonal relations,instrumental role functioning,intrapsychic functioning,and use of objects and participation.The Rosenberg Self-Esteem Scale (RSES,Rosenbeg,1965) were used as a indicator of an attitude of being good enough on 10 items

CONTACTS AND LOCATIONS:
Overall Officials: Gemma Garrido Garcia, Principal Investigator — Consorci Sanitari de Terrassa
Locations (1):
- Consorci Sanitari de Terrassa, Terrassa, Barcelona, Spain

REFERENCES:
- [Background] Wykes T, Reeder C, Landau S, Everitt B, Knapp M, Patel A, Romeo R. Cognitive remediation therapy in schizophrenia: randomised controlled trial. Br J Psychiatry. 2007 May;190:421-7. doi: 10.1192/bjp.bp.106.026575. PMID 17470957
- [Background] Grynszpan O, Perbal S, Pelissolo A, Fossati P, Jouvent R, Dubal S, Perez-Diaz F. Efficacy and specificity of computer-assisted cognitive remediation in schizophrenia: a meta-analytical study. Psychol Med. 2011 Jan;41(1):163-73. doi: 10.1017/S0033291710000607. Epub 2010 Apr 12. PMID 20380784